CLINICAL TRIAL: NCT04616339
Title: A 2-PART, PHASE 1, OPEN LABEL STUDY WITH A 4-PERIOD, 4-SEQUENCE, CROSSOVER DESIGN IN COHORT 1 AND A 2-PERIOD, 2-SEQUENCE CROSSOVER DESIGN IN COHORT 2 TO COMPARE THE SINGLE DOSE PHARMACOKINETICS OF FIVE DIFFERENT FORMULATIONS OF PF-06882961 ADMINISTERED ORALLY TO OTHERWISE HEALTHY ADULT PARTICIPANTS WHO ARE OVERWEIGHT OR HAVE OBESITY
Brief Title: STUDY TO COMPARE PHARMACOKINETICS (PK) OF SINGLE ORAL DOSES OF DIFFERENT PF-06882961 FORMULATIONS IN PARTICIPANTS WHO ARE OVERWEIGHT OR HAVE OBESITY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C3421010; 2020-001016-24 (EudraCT Number)
Record Dates: First submitted 2020-10-30; First posted 2020-11-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Overweight and/or Obesity
MeSH Terms: interventions — danuglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Formulation A (Cohort 1) (Active Comparator): Following an overnight fast of at least 10 hours, subjects received PF-06882961 (Danuglipron) 100 mg immediate release tablet as formulation A at approximately 0800 hours (±2 hours). A minimum of 72 hours between the single 100 mg doses administered in each period was employed
  Interventions: Drug: PF-06882961 100 mg
- Formulation B (Cohort 1) (Experimental): Following an overnight fast of at least 10 hours, subjects received PF-06882961 (Danuglipron) 100 mg immediate release tablet as formulation B at approximately 0800 hours (±2 hours). A minimum of 72 hours between the single 100 mg doses administered in each period was employed
  Interventions: Drug: PF-06882961 100 mg
- Formulation C (Cohort 1) (Experimental): Following an overnight fast of at least 10 hours, subjects received PF-06882961 (Danuglipron) 100 mg immediate release tablet as formulation C at approximately 0800 hours (±2 hours). A minimum of 72 hours between the single 100 mg doses administered in each period was employed
  Interventions: Drug: PF-06882961 100 mg
- Formulation D (Cohort 1) (Experimental): Following an overnight fast of at least 10 hours, subjects received PF-06882961 (Danuglipron) 100 mg immediate release tablet as formulation D at approximately 0800 hours (±2 hours). A minimum of 72 hours between the single 100 mg doses administered in each period was employed
  Interventions: Drug: PF-06882961 100 mg
- Formulation A (Cohort 2) (Active Comparator): Following an overnight fast of at least 10 hours, subjects received PF-06882961 (Danuglipron) 100 mg immediate release tablet as formulation A at approximately 0800 hours (±2 hours). A minimum of 72 hours between the single 100 mg doses administered in each period was employed
  Interventions: Drug: PF-06882961 100 mg
- Formulation E (Cohort 2) (Experimental): Following an overnight fast of at least 10 hours, subjects received PF-06882961 (Danuglipron) 100 mg immediate release tablet as formulation E at approximately 0800 hours (±2 hours). A minimum of 72 hours between the single 100 mg doses administered in each period was employed
  Interventions: Drug: PF-06882961 100 mg

INTERVENTIONS:
Drug: PF-06882961 100 mg — PF-06882961 100 mg will be provided in 5 different oral formulations A, B, C, D, and E. Cohort 1 is a randomized, open-label, single dose, 4-period, 4-sequence, crossover design where the first 2 periods are cross-over (Formulations A and B) and the second 2 periods are crossover (Formulations C and D).
  Cohort 2 is a randomized, open-label, single dose, 2-period, 2 sequence, crossover design (Formulations A and E)

SUMMARY:
The purpose of the study is to evaluate the effect of formulation on relative bioavailability of PF-06882961.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the ICD.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vitals and ECGs. Participants with obesity that are otherwise healthy may be enrolled in this study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* A total body weight >50 kg (110 lb) and BMI of 25.0 to 40.0 kg/m2 at the screening visit.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HBsAg, HBsAb, HBcAb, HCVAb or HIV. Hepatitis B vaccination is allowed.
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2), or participants with suspected MTC per the investigator's judgement.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 halflives (whichever is longer) prior to the first dose of study intervention.
* Use of hormone replacement therapy or oral/injectable contraceptives.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* Participants with known prior participation (ie, randomized and received at least 1 dose of investigational product) in a study involving PF 06882961.
* A positive urine drug test.
* Using a properly sized and calibrated BP cuff, screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.25 × upper limit of normal (ULN);
  * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
  * HbA1c ≥6.5%;
  * Fasting blood glucose ≥126 mg/dL (7 mmol/L);
  * Calcitonin > ULN;
  * eGFR <60 mL/min/1.73 m2 as calculated by the CKD-EPI equation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for Formulations A and B cohort 1 | Day 1 hour (hr) 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48 and end of study (Day 28)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Formulations A and B cohort 1 | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48
Maximum Observed Plasma Concentration (Cmax) for Formulations A and B cohort 1 | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for Formulations A and E cohort 2 | Day 1 hour (hr) 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36, Day 3 hr 48 and end of study (Day 28)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Formulations A and E cohort 2 | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48
Maximum Observed Plasma Concentration (Cmax) for Formulations A and E cohort 2 | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48

SECONDARY OUTCOMES:
Number of Subjects Reporting Treatment-emergent adverse events (AEs) | Baseline through End of Study(Day 28)
Number of Participants With Clinical Laboratory Abnormalities | Baseline, Day 1 and Day 3
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline, Day 1 and Day 3
Number of Participants With Abnormal Electrocardiogram (ECG) | Baseline, Day 1 and Day 3
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for Formulations C and D | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Formulations C and D | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48
Maximum Observed Plasma Concentration (Cmax) for Formulations C and D | Day 1 hr 0, 1, 2, 3, 4, 6, 8, 10, 12, 16, Day 2 hr 24 and 36 and Day 3 hr 48

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421010